CLINICAL TRIAL: NCT00895375
Title: Prevalence of Sleep Disturbances in Psoriasis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00008291
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Psoriasis
Keywords: Dermatology; Skin; Psoriasis; Sleep; Wake Forest; Insomnia
MeSH Terms: conditions — Psoriasis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis patients: 40 subjects (male or female) age 18 or older with psoriasis covering >10% BSA and without a diagnosis of depression.
- Patients without psoriasis: 40 subjects without psoriasis matched for age, sex and BMI, as a control population.

SUMMARY:
The purpose of this study is to compare the sleep quality of patients with psoriasis to patients without psoriasis.

DETAILED DESCRIPTION:
In psoriasis, the burden of disease extends well beyond physical manifestations and can be associated with significant physical, social and psychological impairments. The impact of psoriasis on quality of life has been extensively investigated and demonstrates a negative affect on activities of daily living including sleep. Sleep abnormalities have also been reported in other dermatologic diseases including atopic dermatitis. However, there is relatively little data on the impact of psoriasis on sleep quality and what factors are likely to cause sleep disturbances. Obtaining this information is important because both psoriasis and sleep disorders are associated with cardiovascular disease. A better understanding of sleep problems in psoriasis may help to further our knowledge of psoriasis co-morbidities.

Certain factors associated with psoriasis, including pruritus, depression, and sleep-disordered breathing (obstructive sleep apnea) can independently affect sleep. It would be of particular interest to assess the effect of these factors on sleep quality in psoriasis subjects and the control group to determine what type of sleep problems exist among patients with psoriasis.

This study involves the use of six questionnaires to be given to subjects with psoriasis covering >10% BSA and 40 subjects without psoriasis matched for age, gender and BMI, as a control population. The questionnaires will be given to subjects when they come for their scheduled appointments. The surveys will be completed anonymously and will be collected by a staff member when they are done. A physician will determine the participants' disease severity using the Psoriasis Area and Severity Index (PASI) and will attach the score to their questionnaire.

The questionnaires will cover sleep quality, depression, pruritis, insomnia, hypersomnia, and sleep-disordered breathing. Subjects will be given standard instructions to follow written directions on each questionnaire and will be given an unlimited amount of time to complete the surveys.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis (at least 6 months)

Exclusion Criteria:

* Active depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Wake Forest University Physicians outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Measured prevalence of poor sleep quality in psoriasis subjects as compared to sex-, age-, and BMI-matched subjects without psoriasis, defined as the control population, will be assessed by the Pittsburgh Sleep Quality Index (PSQI). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, PhD, Principal Investigator — Department of Dermatology, Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Dermatology, Winston-Salem, North Carolina, United States